CLINICAL TRIAL: NCT01945086
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group Study of Ustekinumab in Adult Japanese Subjects With Severe Atopic Dermatitis
Brief Title: A Study of Ustekinumab (STELARA®) in Adult Japanese Participants With Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR102538
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, Atopic; Eczema; Ustekinumab; CNTO1275; STELARA
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ustekinumab 45 mg (Experimental)
  Interventions: Drug: Ustekinumab; Other: Concomitant topical medications for atopic dermatitis
- Ustekinumab 90 mg (Experimental)
  Interventions: Drug: Ustekinumab; Other: Concomitant topical medications for atopic dermatitis
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Concomitant topical medications for atopic dermatitis

INTERVENTIONS:
Drug: Ustekinumab — Participants will receive subcutaneous (SC) injections of either ustekinumab 45 mg or ustekinumab 90 mg at Week 0 and Week 4.
  Arms: Ustekinumab 45 mg; Ustekinumab 90 mg
Drug: Placebo — Participants will receive SC injections of placebo at Week 0 and Week 4.
  Arms: Placebo
Other: Concomitant topical medications for atopic dermatitis — Concomitant topical medications (as defined in the protocol) can be used from 4 weeks prior to randomization and throughout the study. However, the dosage cannot be increased and new medications cannot be added until after Week 12.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of 2 doses of ustekinumab compared with placebo (inactive medication) in adult Japanese participants with severe atopic dermatitis.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), placebo-controlled (one of the study medications is inactive), multicenter, parallel group study (each participant group receives different treatments simultaneously). Participants will be randomly assigned in a 1:1:1 ratio to receive either ustekinumab 45 mg, ustekinumab 90 mg, or placebo. The study will consist of a screening period, a 12-week double-blind treatment period, and a 12-week follow-up period. During the double-blind treatment period, participants will receive one subcutaneous injection of study medication at Week 0 and Week 4. Participants will return to the study center for 7 evaluation visits on Weeks 2, 4, 8, 12, 16, 20, and 24. Clinical response will be evaluated by Eczema Area and Severity Index (EASI), Investigator's Global Assessment (IGA), photography, and Dermatology Life Quality Index (DLQI). Participants will record their itch condition twice daily using the participant daily diary from 2 weeks prior to randomization until Week 12. Blood samples will be drawn at time periods during the screening, double-blind treatment, and follow-up periods. Participant safety will be monitored throughout the study. Participants are permitted to use concomitant topical medications, as defined in the protocol and without any increase in dose, from 4 weeks prior to randomization through to the end of the treatment period. After Week 12, additional treatment can be started or the dose of concomitant medications can be increased, if no improvement in clinical response is observed; in these cases EASI, IGA, and photography evaluations will be stopped. The study duration for each participant is expected to be approximately 30 weeks. Ustekinumab (also known as STELARA) is an antibody medication that inhibits the inflammatory proteins IL-12 and IL-23 and is approved as a treatment for moderate to severe plaque-type psoriasis; this study will examine whether ustekinumab can provide benefit in atopic dermatitis and assess for any risks or side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must be Japanese
* Must have a diagnosis of atopic dermatitis, with childhood onset (under age of 13), in accordance with the definition and diagnostic criteria of the Japanese Dermatological Association and must have pruritus and eczematous changes; the condition must be chronic or chronically relapsing in nature
* Inadequate response to, or not willing to use strong treatment with a topical corticosteroid and/or a topical calcineurin inhibitor and/or phototherapy
* Must meet all the following criteria regarding severity of atopic dermatitis: Rajka-Langeland score of 8 to 9; severe or very severe disease as defined in standard treatment guidelines; an Eczema Area and Severity Index (EASI) score of >= 12; and an Investigator's Global Assessment (IGA) score of severe disease or very severe disease
* Must conform to the following tuberculosis (TB) screening criteria: no history of latent or active TB prior to screening; no signs or symptoms suggestive of active TB; no recent close contact with a person with active TB; and a negative Interferon Gamma Release Assay (IGRA) result within 2 months prior to the first administration of study drug

Exclusion Criteria:

* History of or current clinically significant medical illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Has an indeterminate initial and repeat IGRA result or a newly positive IGRA result and is unwilling or unable to undergo TB prophylaxis treatment
* Has received any of the following medications or therapies within 4 weeks prior to randomization: systemic non-steroid immunosuppressive or immunomodulatory drugs; systemic corticosteroids; high daily dose of inhaled corticosteroids; topical corticosteroids of strongest potency for atopic dermatitis; topical antihistamines (including topical doxepin); topical anesthetics; topical nonsteroidal anti-inflammatory drugs; topical counter-irritants (eg, capsaicin, menthol, wintergreen oil); antidepressants or antipsychotics; soporifics; phototherapy including ultraviolet A , ultraviolet B, and psoralen with ultraviolet A (PUVA); hyposensitization (desensitization) therapy
* Has changed the dose and dosing regimen within 4 weeks prior to randomization of any of the following drugs: topical corticosteroid (excluding the strongest potency) for atopic dermatitis; topical calcineurin inhibitor; emollients; anti-leukotriene therapies (including therapies for other allergic indications); systemic histamine H1 blocker (including sleep medications with antihistamine properties); sodium cromoglicate; suplatast tosilate; tranilast; thromboxane A2 inhibitors; and topical or oral herbal preparations for the treatment of atopic dermatitis
* Has received any of the following biologic agents within the following time periods: any marketed immunomodulatory biologic within a period of 3 months or 5 half-lives, whichever is longer, prior to randomization; a biologic agent targeting IL-12 or IL-23, including but not limited to ustekinumab (CNTO 1275), briakinumab (ABT-874), guselkumab (CNTO 1959) or MK-3222 at any point in time; or an experimental biologic therapy within the previous 6 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (13):
- Japan (13):
  - Chitose
  - Habikino
  - Hamamatsu
  - Hiroshima
  - Kumamoto
  - Kurume
  - Kyoto
  - Maebashi
  - Nagasaki
  - Osaka
  - Sapporo
  - Suita
  - Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received subcutaneous (SC) injections of placebo at Week 0 and Week 4.
- Ustekinumab 45 mg: Participants received subcutaneous (SC) injections of ustekinumab 45 milligram (mg) at Week 0 and Week 4.
- Ustekinumab 90 mg: Participants received subcutaneous (SC) injections of ustekinumab 90 mg at Week 0 and Week 4.
Period: Overall Study
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Started | 27 | 24 | 28
Completed | 26 | 24 | 26
Not Completed | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | Total
Number analyzed (Participants) | 27 | 24 | 28 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (10.05) | 37.5 (8.77) | 33.0 (8.85) | 34.2 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 9 | 24
  Male | 19 | 17 | 19 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Eczema Area Severity Index (EASI) Total Score From Baseline at Week 12
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) on a scale of 0 (none) to 3 (severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no eruption) to 6 (greater than [>] 90 percent [%]-100% eruption). The total score is the sum of the four body-region scores, maximum=72, minimum=0, with higher scores reflecting greater disease severity. The total qualitative score is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant and summed to yield the EASI score.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS) included all randomized participants with at least 1 study agent administration irrespective of whether the participant received the assigned treatment, and had at least 1 postdose EASI assessment. Last Observation Carried Forward (LOCF) method was used to impute the missing data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
percent change | -37.54 (37.592) | -38.62 (32.684) | -39.39 (38.710)

2. Secondary Outcome: Number of Participants With an Investigator's Global Assessment (IGA) Score of "Clear" or "Almost Clear" at Week 12
Description: The IGA utilizes a 6-point scale ranging from 0 (clear) to 5 (very severe disease) where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe and 5 (very severe disease).
Time Frame: Week 12
Population: FAS included all randomized participants with at least 1 study agent administration irrespective of whether the participant received the assigned treatment, and had at least 1 postdose EASI assessment. LOCF method was used to impute the missing data.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
participants | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Atopic Dermatitis Itch Scale (ADIS) at Week 12
Description: The atopic dermatitis itch scale (ADIS) will be used to assess pruritus (itching) among participants with AD. It will be evaluated by participant diary kept twice daily,in the morning(morning daily score[MDS]) and evening (Evening Daily Score[EDS]). The start-of-day item set consists of 4 items:itching at time of completing morning diary(Q1),presence of itching during night before(Q2), itching at its worst at night (Q3), and impact of itching on sleep at night(Q4). Appropriate items are summed to yield total score ranging from 0=minimum to 23=maximum, with higher scores reflecting greater itching. The end-of day item set also consists of 4 items: itching at time of completing the evening diary(Q1),the presence of itching during the day(Q2),itching at its worst during the day(Q3),and amount of time the participant experienced eczema-related itching(Q4). Appropriate items are summed to yield total score ranging from 0=minimum to 24=maximum,with higher scores reflecting greater itching.
Time Frame: Baseline and Week 12
Population: FAS population was used for analysis. LOCF method was used to impute the missing data. 'N' (Number of Participants Analyzed) signifies number of participants who were evaluable for this outcome measure. 'n' signifies number of participants who were evaluable at each specific time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
units on a scale
  Baseline (MDS [n=27, 24, 28]) | 8.97 (3.784) | 10.03 (4.615) | 8.71 (3.752)
  Change at Week 12 (MDS [n=27, 24, 28]) | -1.58 (3.030) | -1.68 (3.286) | -2.59 (3.716)
  Baseline (EDS [n=27, 23, 28]) | 10.43 (3.569) | 11.22 (4.371) | 9.45 (3.697)
  Change at Week 12 (EDS [n=27, 23, 28]) | -2.07 (2.624) | -1.91 (3.253) | -2.14 (4.517)

4. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 12
Description: The DLQI is a dermatology-specific quality of life (QOL) instrument designed to assess impact of disease on a participants QOL. It is a 10-item questionnaire that, in addition to evaluating overall, QOL can be used to assess 6 different aspects: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships and treatment. Questions scored on a 4-point Likert scale: 0 (not relevant), 1 (a little), 2 (a lot), and 3 (very much). Scores of individual items (0-3) were added to yield a total score (0-30); higher score = greater impairment of participants QOL.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
units on a scale
  Baseline | 6.3 (3.74) | 6.4 (4.58) | 6.6 (3.74)
  Change at Week 12 | -0.6 (3.96) | -1.7 (3.48) | -1.7 (4.56)

5. Secondary Outcome: Number of Participants With Greater Than or Equal to (>=) 50 Percent (%) and >=75% Decrease in EASI Total Score From Baseline
Description: The EASI score was used to measure the severity and extent of AD and measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) on a scale of 0 (none) to 3 (severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no eruption) to 6 (greater than [>] 90%-100% eruption). The total score is the sum of the four body-region scores, maximum=72, minimum=0, with higher scores reflecting greater disease severity. The total qualitative score is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant and summed to yield the EASI score.
Time Frame: Week 2, 4, 8, 12, 16, 20 and 24
Population: FAS population was used for analysis. 'N' (Number of Participants Analyzed) signifies number of participants who were evaluable for this outcome measure. 'n' signifies number of participants who were evaluable at each specific time point for each arm respectively.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
participants
  Week 2:>=50% Decrease (n=27,24,28) | 3 | 2 | 7
  Week 2:>=75% Decrease (n=27,24,28) | 1 | 0 | 0
  Week 4:>=50% Decrease (n=27,24,27) | 7 | 2 | 9
  Week 4:>=75% Decrease (n=27,24,27) | 2 | 0 | 2
  Week 8:>=50% Decrease (n=27,24,27) | 10 | 5 | 10
  Week 8:>=75% Decrease (n=27,24,27) | 5 | 1 | 3
  Week 12:>=50% Decrease (n=27,24,27) | 11 | 9 | 10
  Week 12:>=75% Decrease (n=27,24,27) | 4 | 2 | 5
  Week 16:>=50% Decrease (n=26,24,27) | 11 | 10 | 12
  Week 16:>=75% Decrease (n=26,24,27) | 5 | 4 | 3
  Week 20:>=50% Decrease (n=26,24,26) | 12 | 8 | 12
  Week 20:>=75% Decrease (n=26,24,26) | 6 | 3 | 5
  Week 24:>=50% Decrease (n=26,24,27) | 8 | 8 | 12
  Week 24:>=75% Decrease (n=26,24,27) | 4 | 4 | 5

6. Secondary Outcome: Number of Participants With an IGA Score of "Clear" or "Almost Clear"
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
participants
  Baseline (n=27, 24, 28) | 0 | 0 | 0
  Week 2 (n=27, 24, 28) | 0 | 0 | 0
  Week 4 (n=27, 24, 27) | 0 | 0 | 0
  Week 8 (n=27, 24, 27) | 0 | 0 | 1
  Week 12 (n=27, 24, 27) | 0 | 0 | 0
  Week 16 (n=26, 24, 27) | 2 | 0 | 1
  Week 20 (n=26, 24, 26) | 2 | 0 | 1
  Week 24 (n=26, 24, 27) | 1 | 0 | 1

7. Secondary Outcome: Number of Participants With Greater Than or Equal to 2 Points Decrease in IGA From Baseline
Description: as for outcome 2
Time Frame: Week 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
participants
  Week 2 (n=27, 24, 28) | 2 | 1 | 4
  Week 4 (n=27, 24, 27) | 5 | 2 | 3
  Week 8 (n=27, 24, 27) | 7 | 3 | 7
  Week 12 (n=27, 24, 27) | 7 | 7 | 7
  Week 16 (n=26, 24, 27) | 6 | 5 | 7
  Week 20 (n=26, 24, 26) | 6 | 6 | 7
  Week 24 (n=26, 24, 27) | 3 | 4 | 6

8. Secondary Outcome: Number of Participants in IGA
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
participants
  Baseline: Clear (n=27,24,28) | 0 | 0 | 0
  Baseline: Almost clear (n=27,24,28) | 0 | 0 | 0
  Baseline: Mild disease (n=27,24,28) | 0 | 0 | 0
  Baseline: Moderate disease (n=27,24,28) | 0 | 0 | 0
  Baseline: Severe disease (n=27,24,28) | 22 | 21 | 24
  Baseline: Very severe disease (n=27,24,28) | 5 | 3 | 4
  Week 2: Clear (n=27,24,28) | 0 | 0 | 0
  Week 2: Almost clear (n=27,24,28) | 0 | 0 | 0
  Week 2: Mild disease (n=27,24,28) | 1 | 0 | 4
  Week 2: Moderate disease (n=27,24,28) | 8 | 5 | 7
  Week 2: Severe disease (n=27,24,28) | 16 | 16 | 16
  Week 2: Very severe disease (n=27,24,28) | 2 | 3 | 1
  Week 4: Clear (n=27,24,27) | 0 | 0 | 0
  Week 4: Almost clear (n=27,24,27) | 0 | 0 | 0
  Week 4: Mild disease (n=27,24,27) | 2 | 0 | 2
  Week 4: Moderate disease (n=27,24,27) | 11 | 8 | 11
  Week 4: Severe disease (n=27,24,27) | 13 | 15 | 12
  Week 4: Very severe disease (n=27,24,27) | 1 | 1 | 2
  Week 8: Clear (n=27,24,27) | 0 | 0 | 0
  Week 8: Almost clear (n=27,24,27) | 0 | 0 | 1
  Week 8: Mild disease (n=27,24,27) | 6 | 1 | 4
  Week 8: Moderate disease (n=27,24,27) | 10 | 12 | 11
  Week 8: Severe disease (n=27,24,27) | 10 | 10 | 8
  Week 8: Very severe disease (n=27,24,27) | 1 | 1 | 3
  Week 12: Clear (n=27,24,27) | 0 | 0 | 0
  Week 12: Almost clear (n=27,24,27) | 0 | 0 | 0
  Week 12: Mild disease (n=27,24,27) | 6 | 5 | 6
  Week 12: Moderate disease (n=27,24,27) | 10 | 8 | 11
  Week 12: Severe disease (n=27,24,27) | 10 | 9 | 7
  Week 12: Very severe disease (n=27,24,27) | 1 | 2 | 3
  Week 16: Clear (n=26,24,27) | 0 | 0 | 0
  Week 16: Almost clear (n=26,24,27) | 2 | 0 | 1
  Week 16: Mild disease (n=26,24,27) | 3 | 3 | 5
  Week 16: Moderate disease (n=26,24,27) | 9 | 9 | 12
  Week 16: Severe disease (n=26,24,27) | 11 | 10 | 6
  Week 16: Very severe disease (n=26,24,27) | 1 | 2 | 3
  Week 20: Clear (n=26,24,26) | 0 | 0 | 0
  Week 20: Almost clear (n=26,24,26) | 2 | 0 | 1
  Week 20: Mild disease (n=26,24,26) | 3 | 3 | 5
  Week 20: Moderate disease (n=26,24,26) | 9 | 9 | 12
  Week 20: Severe disease (n=26,24,26) | 11 | 10 | 6
  Week 20: Very severe disease (n=26,24,26) | 2 | 2 | 2
  Week 24: Clear (n=26,24,27) | 0 | 0 | 0
  Week 24: Almost clear (n=26,24,27) | 2 | 0 | 1
  Week 24: Mild disease (n=26,24,27) | 1 | 4 | 6
  Week 24: Moderate disease (n=26,24,27) | 9 | 7 | 10
  Week 24: Severe disease (n=26,24,27) | 12 | 10 | 8
  Week 24: Very severe disease (n=26,24,27) | 2 | 3 | 2

9. Secondary Outcome: Percent Change From Baseline in EASI Total Score
Description: as for outcome 5
Time Frame: Week 2, 4, 8, 12, 16, 20 and 24
Population: FAS population was used for analysis. 'N' (Number of Participants Analyzed) signifies number of participants who were evaluable for this outcome measure. 'n' signifies number of participants who were evaluable at each specific time point for each arm respectively. LOCF method was not applied to impute the missing data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
percent change
  Week 2 (n=27,24,28) | -24.29 (25.402) | -13.85 (21.391) | -25.72 (24.728)
  Week 4 (n=27,24,27) | -31.69 (28.936) | -21.13 (24.097) | -29.19 (30.409)
  Week 8 (n=27,24,27) | -36.06 (35.840) | -31.15 (28.012) | -34.49 (38.857)
  Week 12 (n=27,24,27) | -37.54 (37.592) | -38.62 (32.684) | -40.84 (38.655)
  Week 16 (n=26,24,27) | -39.97 (40.572) | -38.43 (34.202) | -44.39 (40.154)
  Week 20 (n=26,24,26) | -41.03 (43.495) | -40.59 (31.666) | -46.24 (41.817)
  Week 24 (n=26,24,27) | -35.93 (40.524) | -38.83 (35.697) | -46.19 (41.791)

10. Secondary Outcome: Percent Change From Baseline in EASI Sign of Disease Components
Description: as for outcome 5
Time Frame: Week 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
percent change
  Week 2: Erythema (n=27,24,28) | -19.51 (21.533) | -12.03 (13.049) | -19.13 (19.091)
  Week 4: Erythema (n=27,24,27) | -23.24 (25.710) | -17.17 (15.346) | -21.51 (16.334)
  Week 8: Erythema (n=27,24,27) | -29.19 (27.937) | -24.13 (18.549) | -25.38 (21.390)
  Week 12: Erythema (n=27,24,27) | -30.06 (29.751) | -29.73 (25.421) | -29.89 (21.895)
  Week 16: Erythema (n=26,24,27) | -32.36 (32.911) | -28.36 (30.209) | -34.57 (21.759)
  Week 20: Erythema (n=26,24,26) | -31.81 (31.413) | -32.43 (26.550) | -34.84 (23.922)
  Week 24: Erythema (n=26,24,27) | -28.37 (30.243) | -28.65 (27.249) | -37.25 (23.711)
  Week 2: Induration (n=27,24,28) | -11.99 (34.591) | -12.32 (14.315) | -22.17 (24.515)
  Week 4: Induration (n=27,24,27) | -15.82 (39.898) | -16.58 (17.491) | -24.96 (26.132)
  Week 8: Induration (n=27,24,27) | -19.80 (43.965) | -24.16 (22.658) | -26.98 (29.825)
  Week 12: Induration (n=27,24,27) | -21.23 (49.075) | -26.78 (29.282) | -35.42 (29.943)
  Week 16: Induration (n=26,24,27) | -24.34 (51.739) | -25.82 (32.690) | -38.98 (26.767)
  Week 20: Induration (n=26,24,26) | -27.89 (53.568) | -27.21 (29.162) | -40.58 (31.136)
  Week 24: Induration (n=26,24,27) | -22.45 (50.002) | -26.71 (31.240) | -40.06 (30.864)
  Week 2: Excoriation (n=27,23,28) | -20.65 (21.825) | -11.82 (19.872) | -23.91 (25.419)
  Week 4: Excoriation (n=27,23,27) | -26.38 (28.258) | -18.40 (19.323) | -29.73 (28.764)
  Week 8: Excoriation (n=27,23,27) | -30.56 (35.800) | -25.58 (27.607) | -35.02 (30.400)
  Week 12: Excoriation (n=27,23,27) | -31.29 (37.259) | -30.66 (36.517) | -38.33 (27.953)
  Week 16: Excoriation (n=26,23,27) | -33.11 (40.899) | -25.50 (41.929) | -44.25 (27.690)
  Week 20: Excoriation (n=26,23,26) | -33.23 (42.648) | -23.55 (36.947) | -40.67 (33.036)
  Week 24: Excoriation (n=26,23,27) | -26.40 (37.853) | -22.74 (37.555) | -42.07 (33.992)
  Week 2: Lichenification (n=267,24,28) | -14.90 (20.292) | -8.46 (16.879) | -15.87 (18.500)
  Week 4: Lichenification(n=27,24,27) | -23.38 (25.947) | -10.21 (23.359) | -20.24 (24.284)
  Week 8: Lichenification (n=27,24,27) | -26.52 (28.515) | -19.40 (22.871) | -28.07 (27.887)
  Week 12: Lichenification (n=27,24,27) | -28.62 (31.241) | -24.36 (29.272) | -33.06 (25.443)
  Week 16: Lichenification (n=26,24,27) | -32.64 (34.378) | -22.18 (34.489) | -37.47 (27.046)
  Week 20: Lichenification (n=26,24,26) | -33.24 (35.094) | -23.36 (43.750) | -41.71 (30.241)
  Week 24: Lichenification (n=26,24,27) | -32.05 (33.470) | -20.96 (45.278) | -40.19 (26.696)

11. Secondary Outcome: Percent Change From Baseline of Body Region Scores in EASI
Description: as for outcome 5
Time Frame: Week 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
percent change
  Week 2: Head/neck (n=27,24,28) | -20.28 (22.410) | -6.97 (24.488) | -29.50 (9.492)
  Week 4: Head/neck (n=27,24,27) | -26.22 (36.637) | -17.46 (25.632) | -34.15 (32.087)
  Week 8: Head/neck (n=27,24,27) | -29.34 (64.066) | -34.27 (27.380) | -38.65 (28.580)
  Week 12: Head/neck (n=27,24,27) | -32.82 (52.925) | -36.28 (39.256) | -45.34 (25.282)
  Week 16: Head/neck (n=26,24,27) | -37.27 (58.582) | -38.31 (37.155) | -52.12 (23.578)
  Week 20: Head/neck (n=26,24,26) | -35.20 (59.298) | -42.63 (38.094) | -46.30 (35.652)
  Week 24: Head/neck (n=26,24,27) | -24.84 (89.446) | -37.20 (39.828) | -49.63 (28.510)
  Week 2: Upper limbs (n=27,24,28) | -26.64 (29.149) | -14.47 (22.285) | -28.53 (26.760)
  Week 4: Upper limbs (n=27,24,27) | -33.25 (38.613) | -21.62 (23.746) | -30.26 (29.646)
  Week 8: Upper limbs (n=27,24,27) | -44.58 (38.100) | -32.57 (28.600) | -38.11 (37.205)
  Week 12: Upper limbs (n=27,24,27) | -40.64 (42.146) | -36.55 (35.946) | -47.01 (39.135)
  Week 16: Upper limbs (n=26,24,27) | -42.01 (45.743) | -32.55 (47.614) | -42.94 (42.543)
  Week 20: Upper limbs (n=26,24,26) | -41.48 (46.700) | -37.71 (36.660) | -48.20 (37.501)
  Week 24: Upper limbs (n=26,24,27) | -39.61 (45.005) | -39.36 (36.535) | -50.89 (39.446)
  Week 2: Trunk (n=27,24,28) | -27.82 (27.633) | -18.16 (22.783) | -21.84 (33.368)
  Week 4: Trunk (n=27,24,27) | -34.42 (34.730) | -20.59 (26.028) | -23.51 (46.987)
  Week 8: Trunk (n=27,24,27) | -32.28 (49.544) | -27.99 (29.551) | -29.26 (54.157)
  Week 12: Trunk (n=27,24,27) | -33.38 (57.021) | -36.89 (35.351) | -31.65 (54.961)
  Week 16: Trunk (n=26,24,27) | -35.33 (59.694) | -28.96 (41.260) | -37.87 (54.763)
  Week 20: Trunk (n=26,24,26) | -36.37 (62.253) | -32.68 (36.306) | -41.92 (58.260)
  Week 24: Trunk (n=26,24,27) | -28.39 (59.596) | -31.25 (40.207) | -39.77 (56.008)
  Week 2: Lower limbs (n=27,24,28) | -19.84 (29.862) | -9.17 (32.015) | -26.15 (26.073)
  Week 4: Lower limbs (n=27,24,27) | -26.46 (33.485) | -21.32 (33.541) | -33.12 (37.005)
  Week 8: Lower limbs (n=27,24,27) | -31.23 (46.154) | -31.88 (36.302) | -27.56 (82.889)
  Week 12: Lower limbs (n=27,24,27) | -34.79 (45.961) | -42.01 (35.358) | -32.39 (83.114)
  Week 16: Lower limbs (n=26,24,27) | -36.98 (48.713) | -46.30 (34.942) | -36.87 (84.182)
  Week 20: Lower limbs (n=26,24,26) | -38.06 (53.187) | -45.50 (34.350) | -38.92 (86.354)
  Week 24: Lower limbs (n=26,24,27) | -33.60 (50.984) | -41.55 (40.522) | -39.80 (87.186)

12. Secondary Outcome: Number of Participants With Mild or Absent Key Sign of Atopic Dermatitis (AD)
Description: The EASI score was used to measure the severity and extent of AD and measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) on a scale of 0 to 3 where 0=none, 1=mild, 2=moderate, 3=severe, on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no eruption) to 6 (greater than [>] 90%-100% eruption). The total score is the sum of the four body-region scores, maximum=72, minimum=0, with higher scores reflecting greater disease severity. The total qualitative score is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant and summed to yield the EASI score.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 27 | 24 | 28
participants
  Baseline: Erythema (n=27,24,28) | 0 | 0 | 0
  Week 2: Erythema (n=27,24,28) | 1 | 0 | 1
  Week 4: Erythema (n=27,24,27) | 4 | 0 | 1
  Week 8: Erythema (n=27,24,27) | 4 | 1 | 2
  Week 12: Erythema (n=27,24,27) | 5 | 5 | 3
  Week 16: Erythema (n=26,24,27) | 4 | 4 | 7
  Week 20: Erythema (n=26,24,26) | 4 | 4 | 5
  Week 24: Erythema (n=26,24,27) | 5 | 3 | 6
  Baseline: Induration (n=27,24,28) | 1 | 0 | 0
  Week 2: Induration (n=27,24,28) | 1 | 0 | 2
  Week 4: Induration (n=27,24,27) | 5 | 0 | 3
  Week 8: Induration (n=27,24,27) | 4 | 1 | 3
  Week 12: Induration (n=27,24,27) | 3 | 6 | 7
  Week 16: Induration (n=26,24,27) | 6 | 5 | 8
  Week 20: Induration (n=26,24,26) | 7 | 3 | 7
  Week 24: Induration (n=26,24,27) | 5 | 3 | 8
  Baseline: Excoriation (n=27,24,28) | 0 | 1 | 1
  Week 2: Excoriation (27,24,28) | 2 | 2 | 4
  Week 4: Excoriation (n=27,24,27) | 5 | 2 | 7
  Week 8: Excoriation (n=27,24,27) | 5 | 3 | 7
  Week 12: Excoriation (n=27,24,27) | 4 | 9 | 6
  Week 16: Excoriation (n=26,24,27) | 7 | 7 | 9
  Week 20: Excoriation (n=26,24,26) | 7 | 4 | 7
  Week 24: Excoriation (n=26,24,27) | 4 | 5 | 8
  Baseline: Lichenification (n=27,24,28) | 0 | 1 | 0
  Week 2: Lichenification (n=27,24,28) | 1 | 1 | 2
  Week 4: Lichenification (n=27,24,27) | 4 | 0 | 3
  Week 8: Lichenification (n=27,24,27) | 4 | 2 | 2
  Week 12: Lichenification (n=27,24,27) | 4 | 6 | 5
  Week 16: Lichenification (n=26,24,27) | 6 | 4 | 8
  Week 20: Lichenification (n=26,24,26) | 6 | 4 | 7
  Week 24: Lichenification (n=26,24,27) | 5 | 5 | 7

ADVERSE EVENTS:
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 20/27 | 18/24 | 16/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Ustekinumab 45 mg (N=24) | Ustekinumab 90 mg (N=28)
Nasopharyngitis (Infections and infestations) | 7 | 6 | 6
Impetigo (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Kaposi's varicelliform eruption (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Fatty liver alcoholic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 | 4 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema ab igne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2
Aspartate aminotransferase (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.